CLINICAL TRIAL: NCT02869711
Title: Impact of a Training-action About Projects Leading for the Improvement of Care Quality in Managing Practice of Health Executive
Acronym: ImpactFA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC11.244
Record Dates: First submitted 2016-08-09; First posted 2016-08-17 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Health Care Quality Management (no Condition).

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Health care quality management

SUMMARY:
The present study focuses on the quality of care and how the health executives can bring it to a central place in their management. A training-action has been set-up at the Health Executive training institute (University Hospital Grenoble) to improve care quality. Reports prepared by students (tutored projects) related to operational diagnosis and action plans about care quality improvement are given to health executives. The objective is to evaluate how the health executive will use the tutored project to improve care quality and set-up actions.The hypothesis is that the health executive will use the tutored project to improve project management.

DETAILED DESCRIPTION:
Every year, 9 voluntary health executives will be included and followed during 1 year. The experience will be done 3 times (3 years).

It is a qualitative study using 3 forms to recover data: group focus, individual interviews, project monographs. Speeches coding will enable to test the hypothesis from 2 analysis points: place of health executive and place of tutored project.

The study will be resulting in recommendations to health executives for their management methods and taken into account to define training.

ELIGIBILITY:
Inclusion Criteria:

* The volunteers are health executives with diploma

Exclusion Criteria:

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Health Executive volunteers
Sampling Method: Non-Probability Sample
Enrollment: 27 (Estimated)
Dates: Start 2011-07; Primary Completion 2016-09 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Change in the managerial practices of health executives about health care quality management after tutored projects. | 1 year for each volunteer.
  The subjects are not patients but health executive managers. The study foccuses on their management pratices and changes after tutored projects. There are 2 analysis criteria: place of health executive and place of tutored project.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Philippe DUJARDIN, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital Grenoble, Grenoble, France